

# STATISTICAL AND EPIDEMIOLOGICAL ANALYSIS PLAN (SEAP) FOR NON-INTERVENTIONAL STUDIES (NIS)

| Document Number: | c37922104-02 |
|---|---|
| BI Study Number: | 1245-0201 |
| BI Investigational<br>Product(s) | Jardiance® (empagliflozin) |
| Title: | Statistical and Epidemiological Analysis Plan (SEAP) for Post-<br>authorization safety study (PASS) to assess the risk of acute<br>pancreatitis in type 2 diabetes mellitus (T2DM) patients newly<br>initiating empagliflozin compared to other oral non-incretin/non-<br>sodium glucose co-transporter-2 inhibitors (SGLT2)-based glucose<br>lowering agents |
| Brief lay title: | To assess the risk of acute pancreatitis in patients with type 2 diabetes treated with empagliflozin |
| SEAP version identifier: | 1.0 |
| Date of last version of SEAP: | 03 December 2021 |
| NIS Statistician [SEAP author] | |
| NIS [SEAP reviewer] | Global Epidemiology |
| NIS Data [SEAP reviewer] | |
| Page 1of 27 | |
| Proprietary confidential information © 2022 Boehringer Ingelheim Group of companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission | |

be passed on, reproduced, published of otherwise used without prior written permission


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## **TABLE OF CONTENTS**

| TITLE PA | GE | 1 |
|---|---|---|
| TABLE OI | F CONTENTS | 2 |
| 1. | LIST OF ABBREVIATIONS | 4 |
| 2. | RESPONSIBLE PARTIES | 5 |
| 3. | PURPOSE AND SCOPE | 6 |
| 4. | AMENDMENTS AND UPDATES | 6 |
| 5. | RESEARCH QUESTION AND OBJECTIVE | 6 |
| 6. | RESEARCH METHODS | 6 |
| 6.1 | STUDY DESIGN | 6 |
| 6.2 | SETTING | 6 |
| 6.2.1 | Study period | 6 |
| 6.2.2 | Baseline period (lookback period) | 7 |
| 6.2.3 | Follow up | 7 |
| 6.3 | STUDY POPULATION | 7 |
| 6.4 | STUDY VISITS | 7 |
| 7. | VARIABLES | 8 |
| 7.1 | EXPOSURES | 8 |
| 7.1.1 | Operational definitions on how to identify each of the index medication cohorts: | 8 |
| 7.1.2 | Definition of continuous exposure, discontinuation, switch or add-on | 9 |
| 7.1.3 | Definition the censored follow-up end | 9 |
| 7.2 | OUTCOMES | 10 |
| 7.3 | COVARIATES | 10 |
| 8. | DATA SOURCES | 10 |
| 9. | DATA MANAGEMENT AND SOFTWARE/TOOLS | 10 |
| 9.1 | SOFTWARE/TOOLS | 10 |
| 9.2 | HANDLING OF MISSING VALUES | 11 |
| 9.3 | HANDLING OF INCONSISTENCIES IN DATA AND OUTLIERS | 11 |
| 10. | DATA ANALYSIS | 11 |
| 10.1 | DEFINITIONS | 11 |
| 10.2 | PROPENSITY SCORE | 11 |
| 10.3 | MAIN ANALYSIS | 11 |

c37922104-02

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)


| Proprietary | confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies |
|---|---|
| 10.4 | META-ANALYSIS11 |
| 10.6 | SENSITIVITY ANALYSIS |
| 10.7 | SAFETY ANALYSIS |
| 11. | QUALITY CONTROL |
| 12. | REFERENCES |
| 12.1 | PUBLISHED REFERENCES |
| 12.2 | UNPUBLISHED REFERENCES |
| ANNEX 1. | LIST OF ICD 9 AND ICD 10 CODES FOR COHORT CREATION19 |
| ANNEX 2. | MEDICATION CODES USED TO DEFINE EXPOSURES AND EXCLUSION |
| | CRITERIA OR CENSORING20 |
| ANNEX 3. | STUDY COVARIATES22 |

ANNEX 4. REVIEWERS AND APPROVAL SIGNATURES ......27

c37922104-02

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 1. LIST OF ABBREVIATIONS

BI Boehringer Ingelheim

CI Confidence Interval

DMRP Data management and review plan

HDPS High dimensional propensity score

IHD Instant Health Data

IQR Interquartile range

NIS Non-interventional study

SEAP Statistical and epidemiological analysis plan

SGLT2i Sodium glucose co-transporter-2 inhibitor

T2DM Type 2 diabetes mellitus

US United States


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 2. RESPONSIBLE PARTIES

NIS Statistician [SEAP author]:

| Name, degree(s) | Title | Affiliation | Address |
|-----------------|--------------------------|-------------|---------|
| | Global<br>Epidemiologist | | |

SEAP reviewers are:

| • | BI NIS [SEAP reviewer] (in all cases): Global Epidemiology | |
|---|---|---|
| • | NIS Data [SEAP reviewer] (in all cases): | and |
| • | [SEAP reviewer] (for all globally initiated studies and for local studies) involving BI products and Global NIS not involving BI products: | |
| | , and | |
| • | TSTAT (for NISnd only): Not Applicable | |
| • | TM Epi [SEAP reviewer] (When BI NIS is not TM Epi; in all cases): Global Epidemiology | |

c37922104-02

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 3. PURPOSE AND SCOPE

SEAP reviewers are expected to be familiar with the NIS protocol entitled "Post-authorization safety study (PASS) to assess the risk of acute pancreatitis in type 2 diabetes mellitus (T2DM) patients newly initiating empagliflozin compared to other oral non-incretin/non-sodium glucose co-transporter-2 inhibitors (SGLT2)-based glucose lowering agents", version 1.0 dated 29 November 2021 unless otherwise stated.

The SEAP addresses the details of the implementation of this study. In the SEAP, you can find the detailed operational definitions on how to identify each of the index medication cohorts, detailed data analysis plan such as the propensity score matching, meta-analysis, and Main analysis plan. In addition, the study covariates are captured in the <u>Annex 3</u>.

#### 4. AMENDMENTS AND UPDATES

None.

## 5. RESEARCH QUESTION AND OBJECTIVE

This non-interventional cohort study using data from two large United States claims databases will describe the risk of acute pancreatitis among patients with type 2 diabetes mellitus (T2DM) initiating empagliflozin between from 1 August 2014 to the latest data-cut available in Marketscan (30 September 2020) and Optum (31 March 2021).

#### Primary Objective:

• To compare the incidence rate of acute pancreatitis in T2DM patients initiating empagliflozin to new users of other oral non-incretin/non-SGLT2i-containing glucose lowering drugs between 1 August 2014 and the latest data-cut available in Marketscan (30 September 2020) and Optum (31 March 2021).

#### 6. RESEARCH METHODS

#### 6.1 STUDY DESIGN

Please see the study protocol.

#### 6.2 SETTING

Please see the study protocol.

## 6.2.1 Study period

The patient selection period will be from 01 August 2014 to the latest data-cut available in Marketscan (30 September 2020) and Optum (31 March 2021). Patients will be selected into the study at any time during this period once they fulfil the study eligibility criteria.

c37922104-02

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 6.2.2 Baseline period (lookback period)

Patients are required to have at least 6 months of continuous registration in the database prior to initiation of empagliflozin or a comparator drug. The look-back period is defined as 6 months prior to the index date and including the index date. The look-back period was specified to confirm new medication use (i.e., having a first prescription claim for empagliflozin or other oral non-incretin/non-SGLT2i-based glucose lowering agents without use of these medications in the prior 6 months) and describe baseline parameters, such as prior medical history and medications.

#### 6.2.3 Follow up

Follow up starts at the day after the index date until the first qualifying event has been met (see table 2 and 3 of the study protocol).

#### 6.3 STUDY POPULATION

Please see the study protocol for the details.

Codes to select study population are listed in <u>Annex 1</u>.

One of the risk factors of acute pancreatitis is severity of diabetes and diabetes duration [R10-6620, R10-2088]. In the Optum and Marcketscan databases duration of diabetes can not be measured for all patients, therefore chronic use of insulin at baseline was selected as an exclusion criterion to remove severe cases of diabetes who are already at higher risk of developing acute pancreatitis. We defined 60 (or more) days of continuous exposure as chronic use of insulin for the exclusion criteria.

The operational steps are as follows:

Insulin prescriptions will be extracted during the 6 months baseline period according to insulin medication codes listed in <u>Annex 2</u>. Despite the variations in package size and dosing schedule, a majority of insulin prescriptions are dispensed with 30 days' supply [<u>R21-4257</u>, <u>R21-4258</u>].

The continuous exposure episode of insulin is constructed by linking insulin prescriptions with allowed less or equal 30 gap days [R21-0580]. If any of continuous exposure episodes have 60 or more than 60 days duration, this will be considered as chronic use of insulin and this patient will be excluded from the cohort.

#### 6.4 STUDY VISITS

Not applicable.


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7. VARIABLES

Study variables are explained the study protocol <u>section 9.3</u>. you can find attritional operational definitions below:

#### 7.1 EXPOSURES

Please check section 9.3.1 of the study protocol.

# 7.1.1 Operational definitions on how to identify each of the index medication cohorts:

For index medication determination, we first select all patients with any of Empagliflozin, TZD, SU and Metformin prescriptions within study period. Then we evaluate index drug for each patient following this order: Empagliflozin  $\rightarrow$  TZD  $\rightarrow$  SU  $\rightarrow$  Metformin. Therefore, each patient will be classified into one of index cohorts only once. The details for Empagliflozin initiators are provided below and all other drugs follow the same approach.

#### Empagliflozin initiators:

- 1. Between Aug 2014 and latest data cut we will choose all Empagliflozin new users. The date of first Empagliflozin prescription will be selected as index date. New users should not have any prescriptions for Empagliflozin in 6 months prior to the index date.
- 2. In the next step we will check which of the Empagliflozin initiators use metformin, or SU in the 6-month baseline period



Figure 1 Diagram for Mono, Combo or Triple groups creations

Code list for exposure variables is available in Annex 2.

The index date in both groups will be the date of prescription of empagliflozin or other hypoglycaemic therapies (index medication), and the planned study follow-up period starts at the day after index date.

c37922104-02

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 7.1.2 Definition of continuous exposure, discontinuation, switch or add-on

The continuous exposure periods of index drug have been created by linking all prescriptions with days of supply with 30 days grace period in between. Note: 30 days grace period is used in main analysis. 90 days grace period will be used in sensitivity analysis. The discontinuation is when there is more than 30 days gap from current prescription exposure end to next prescription date. The discontinuation date is 30 days after the end of days of supply of the last prescription date.

Addition of a new medication means when the prescription date of this new medication is before the last prescription date of the index continuous exposure. The prescription date of new medication is add-on date.

Switch to new medication means the prescription date of this new medication is on or after the last prescription date of the index continuous exposure and before the end of discontinuation. The prescription date of new medication is switch date. Different scenarios for switch, discontinue, or add on were mentioned in the study protocol.

#### 7.1.3 Definition the censored follow-up end

The study will be conducted utilizing a modified "as-treated" approach. The follow up time starts from index date till the earliest date of these following events:

- 1. Discontinuation of index drug.
- 2. Switch or add-on the within treatment line comparator (other SGLT2 in empagliflozin group or the comparator group. Please refer to <u>Table 1</u> for different switch or add-on scenarios for each group.
- 3. Outcome: AP event. The first date of AP event is the event date.
- 4. The minimum date of death date or enrollment end date or study end date

As long as it is not the treatment line comparator, patients are allowed to add a non-incretin/non-SGLT2i hypoglycemic agent to their index therapy and can also switch to non-incretin/non-SGLT2i hypoglycemic agents.

Based on the feasibility studies, the patients having fixed dose of Empagliflozin + Metformin are definied as dual Empagliflozin patients. The index date is the first prescription of fixed dose prescription.

For the patients starting Metformin then Empagliflozin, these patients are free dose Empagliflozin + Metformin dual patients and they are definied as dual Empagliflozin patients by following exposure group definition process. The index date is the first Empagliflozin prescription date.

For both situations, the index drug is Empagliflozin. The cencor date will be captured by following the same rule.




Figure 2 Diagram for definition of the censored end of follow up

#### 7.2 OUTCOMES

Please check section 9.3.2. of the study protocol.

#### 7.3 COVARIATES

Please check section 9.3.3. of the study protocol. List of covariates and operational definitions are added to <u>Annex 3</u>.

#### 8. DATA SOURCES

Please check section 9.4 of the study protocol.

#### 9. DATA MANAGEMENT AND SOFTWARE/TOOLS

Data is stored using the secured Instant Health Data (IHD) platform (https://www.bhei.com/product). Access to the data is granted by password to trained, BI personnel only. All study details are addressed either in the protocol, SEAP, or DMRP.

#### 9.1 SOFTWARE/TOOLS

The cohort selection part will be conducted in IHD platform and the data analysis will be run in BI internal server using SAS software 9.4 ( ) or R Studio 3.5.2.

c37922104-02

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.2 HANDLING OF MISSING VALUES

The absence of a code for a condition will be interpreted as an absence of the event. If a study variable is totally missing from a database, it is excluded from the analysis of the pooled data. If a variable is missing for only some of the patients a missing data category will be added and utilized in the analysis.

#### 9.3 HANDLING OF INCONSISTENCIES IN DATA AND OUTLIERS

For lab values, distribution of each variable will be assessed. The extreme outliers will be treated as missing values approaches to handling missing values are described in the previous section.

### 10. DATA ANALYSIS

#### 10.1 **DEFINITIONS**

Please check the study protocol section 9.7.1.

#### 10.2 PROPENSITY SCORE

Please check study protocol section 9.7.2.

#### 10.3 MAIN ANALYSIS

Please check study protocol section 9.7.3.

#### 10.4 META-ANALYSIS

Please check study protocol section 9.7.4.



c37922104-02

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)




c37922104-02

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)


| Proprietary confidential | information © 2022 Boehi | rınger İngelheim İnternatio | onal GmbH or one or more o | of its affiliated companies |
|---|---|---|---|---|

c37922104-02

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

c37922104-02

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 10.6 SENSITIVITY ANALYSIS

See relevant section of the study protocol.

#### 10.7 SAFETY ANALYSIS

Not applicable based on secondary use of data without any potential that any employee of BI or agent working on behalf of BI will access individually identifiable patient data.

### 11. QUALITY CONTROL

The quality control, review, and monitoring plan are summarized below. Greater details are documented in the NIS-DMRP.

All measures created, cohorts developed, statistical analyses implemented, and tables completed will be conducted by two analysts independently. After completing the whole analysis, each analyst will undergo quality control review for the other analyst's work. The final results need to be consistent results from both analysts.

This protocol will be strictly followed in the study. All changes to this protocol will be documented in protocol amendments.

All programs for data management and data analyses written by study statistician(s) will be self-documenting with comments about the data handling process, the population selection and the analysis performed by the program. The documentation will be sufficient for another statistician to be able to repeat the program. A statistician other than the one who writes the program will carry out quality control checks of these programs. The programming quality control (QC) will be performed for all programs related to the database, its individual datasets from different registers and statistical analyses. The QC will be documented with the following information:

- Name of the program
- Purpose of the program
- Name of the programmer
- Validation status and date of validation
- Updates and dates of updates
- Name of the QC statistician
- QC findings or comments
- Date of QC

The statistician responsible for the QC of a program will ensure that:

- The correct dataset and population has been used
- The analysis is carried out according to the SEAP
- The analysis results are consistent

c37922104-02

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- The output is in line with the table shells in the SEAP
- The analysis can be interpreted in both statistical and clinical terms.

All QC findings by the QC statistician will be documented, and corrections are made to the programs accordingly. All changes are documented as updates to the original program.

The raw dataset and statistical programs used for generating the data included in the final study report will be kept in electronic format and be available for auditing and inspection.


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## 12. REFERENCES

#### 12.1 PUBLISHED REFERENCES

| R11-2165 | Schneeweiss S. Sensitivity analysis and external adjustment for unmeasured confounders in epidemiologic database studies of therapeutics. Pharmacoepidemiol Drug Saf 2006; 15; 291-303. |
|---|---|
| R13-3590 | Austin PC. Optimal caliper widths for propensity-score matching when estimating differences in means and differences in proportions in observational studies. Pharm Stat 2011; 10(2); 150-161. |
| R20-3573 | Zhang Z, Kim HJ, Lonjon G, Zhu Y, AME Big-Data Clinical Trial Collaborative Group. Balance diagnostics after propensity score matching. Ann Transl Med 2019; 7(1); 16 |
| R13-0525 | Schneeweiss S, Rassen JA, Glynn RJ, Avorn J, Mogun H, Brookhart MA. High-dimensional propensity score adjustment in studies of treatment effects using health care claims data. Epidemiology 2009; 20(4); 512-522. |
| R13-2767 | Rassen JA, Glynn RJ, Brookhart MA, Schneeweiss S. Covariate selection in high-dimensional propensity score analyses of treatment effects in small samples. Am J Epidemiol 2011; 173(12); 1404-1413. |
| R21-0580 | Hadjiyianni I, Desai U, Suzuki S, Ivanova JI, Cao D, Kirson NY, et al. Basal insulin persistence, associated factors, and outcomes after treatment initiation: a retrospective database study among people with type 2 diabetes mellitus in Japan. Diabetes Ther 2017; 8; 149-166. |
| R21-4257 | Buysman E, Conner C, Aagren M, Bouchard J, Liu F. Adherence and persistence to a regimen of basal insulin in a pre-filled pen compared to vial/syringe in insulin-naive patients with type 2 diabetes. DOI: 10.1185/03007995.2011.598500. Curr Med Res Opin 2011; 27(9); 1709-1717. |
| R21-4258 | Eby EL, Bajpai S, Faries DE, Haynes VS, Lage MJ. The association between adherence to insulin therapy and health care costs for adults with type 2 diabetes: evidence from a U.S. retrospective claims database. DOI: 10.18553/jmcp.2020.26.9.1081. J Managed Care Spec Pharm 2020; 26(9); 1081-1089. |
| R10-6620 | Girman CJ, Kou TD, Cai B, Alexander CM, O'Neill EA, Williams-Herman DE, Katz L. Patients with type 2 diabetes mellitus have higher risk for acute pancreatitis compared with those without diabetes. Diabetes Obes Metab 2010; 12(9); 766-771. |
| R10-2088 | Noel RA, Braun DK, Patterson RE, Bloomgren G. Increased risk of acute pancreatitis and biliary disease observed in patients with type 2 diabetes: a |


| Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies | |
|---|---|
| | retrospective cohort study. Diabetes Care 2009; 32(5); 834-838. |
| R17-2092 | Patorno E, Everett BM, Goldfine AB, Glynn RJ, Liu J, Gopalakrishnan C, et al. Comparative cardiovascular safety of glucagon-like peptide-1 receptor agonists versus other antidiabetic drugs in routine care: a cohort study. Diabetes Obes Metab 2016; 18(8); 755-765. |
| R20-1531 | Anand ER, Major C, Pickering O, Nelson M. Acute pancreatitis in a COVID-19 patient. DOI: 10.1002/bjs.11657. British Journal of Surgery, Online ahead of print, 2020 Apr 27, doi: 10.1002/bjs.11657; 2020. p. e182 |
| R20-1532 | Hadi A, Werge M, Kristiansen KT, Pedersen UG, Karstensen JG, Novovic S, et al. Coronavirus disease-19 (COVID-19) associated with severe acute pancreatitis: case report on three family members. DOI: 10.1016/j.pan.2020.04.021. Pancreatology, Article in Press, Corrected Proof, Available online 5 May 2020, doi: 10.1016/j.pan.2020.04.021; 2020. p. 665-667. |
| R20-1536 | Wang F, Wang H, Fan J, Zhang Y, Wang H, Zhao Q. Pancreatic injury patterns in patients with COVID-19 pneumonia. DOI: 10.1053/ Gastroenterology, Journal Pre-proof, Published online: April 01, 2020, doi: 10.1053/j.gastro.2020.03.055; 2020. p. 367-370. |
| R20-3357 | Liu F, Long X, Zou W, Fang M, Wu W, Li W, et al. Highly ACE2 expression in pancreas may cause pancreas damage after SARS-CoV-2 infection. DOI: 10.1101/2020.02.28.20029181. doi: 10.1101/2020.02.28.20029181; 2020. |
| R21-1729 | Bulthuis MC, Boxhoorn L, Beudel M, Elbers PWG, Kop MPM, Wanrooij RLJ van, et al. Acute pancreatitis in COVID-19 patients: true risk? Source: Scand J Gastroenterol 2021; 56(5); 585-587. |
| R21-1730 | Troncone E, Salvatori S, Sena G, Cristofaro E de, Alfieri N, Marafini I, et al. Low frequency of acute pancreatitis in hospitalized COVID-19 patients. Pancreas 2021; 50(3); 393-398. |
| R14-4775 | Quan H, Sundararajan V, Halfon P, Fong A, Burnand B, Luthi JC, Saunders LD, Beck CA, Feasby TE, Ghali WA. Coding algorithms for defining comorbidities in ICD-9-CM and ICD-10 administrative data. Med Care 2005; 43(11); 1130-1139. |

### 12.2 UNPUBLISHED REFERENCES

Not applicable.

c37922104-02

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# ANNEX 1. LIST OF ICD 9 AND ICD 10 CODES FOR COHORT CREATION

| Condition | ICD 9 codes <sup>1</sup> | ICD 10 codes <sup>2</sup> |
|---|---|---|
| T1DM | 250.X1, 250.X3 | E10.xx |
| T2DM | 250.X0, 250.X2 | E11.xx |
| Gestational diabetes | 648.8x | O24.1x, O24.4x |
| Secondary diabetes | 249.xx | E08.xx, E09.xx,E13.xx |
| Acute pancreatitis | 577.0 | K85.xx |
| Chronic pancreatitis | 577.1 | K86.1 Other chronic pancreatitis |
| Pancreatitis cancer | 157.xx | C25.xx |
| Other disease of pancreatitis | 577.2, 577.8, 577.9 | K86.2, K86.3, K86.8x, K86.9 |

<sup>1. 2015</sup> ICD-9-CM Diagnosis Codes: http://www.icd9data.com/2015/Volume1/default htm accessed at 14 March 2020

001-MCS-90-118 RD-20 (2.0) / Saved on: 03 Feb 2021

<sup>2. 2019</sup> ICD-10-CM Codes: https://www.icd10data.com/ICD10CM/Codes accessed at 14 March 2020


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# ANNEX 2. MEDICATION CODES USED TO DEFINE EXPOSURES AND EXCLUSION CRITERIA OR CENSORING

| Medication Class / Generic (Brand) Name Medication for Evrosum Crowns Definition |
|---|
| Medication for Exposure Groups Definition |
| Empagliflozin |
| Empagliflozin (Jardiance): Empa Mono |
| Empa+ Met |
| Metformin + Empagliflozin (Synjardy): Empa Dual |
| Metformin + Empagliflozin extended-release (Synjardy XR): Empa Dual |
| Metformin |
| Metformin (Glucophage, metformin hydrochloride, Fortamet, Glumetza, Riomet): Metf |
| Mono |
| Met + TZD |
| Metformin + Pioglitazone (Actoplus Met): Metf + TZD |
| Metformin + Rosiglitazone (Avandamet): Metf + TZD |
| Met + SU |
| Metformin + Glipizide (Metaglip): Metformin and SU Dual |
| Metformin + Glyburide (Glucovance): Metformin and SU Dual |
| SU (Combine 1st and 2nd gen) |
| Glimepiride (Amaryl) |
| Glipizide (Glucotrol) |
| Glyburide (DiaBeta) |
| Glynase |
| Glycron |
| Micronase |
| Acetohexamide (Dymelor) |
| Chlorpropamide (Diabinese) |
| Tolazamide (Tolinasel) |
| Tolbutamide (Orinase) |
| TZD |
| Alogliptin + Pioglitazone (Oseni) |
| Pioglitazone (Actos) |
| Rosiglitazone (Avandia) |
| SU+ TZD |
| Glimepiride + Rosiglitazone (Avandaryl) |
| Glimepiride + Pioglitazone (Duetact) |


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies Medicaiton used in exclusion or censoring exposure duration: Dipeptidyl peptidase-4 inhibitor (DPP-4i) Alogliptin (Nesina) Metformin + Alogliptin (Kazano) Linagliptin (Tradjenta) Metformin + Linagliptin (Jentadueto) Empagliflozin + Linagliptin (Glyxambi) Saxagliptin (Onglyza) Metformin + Saxagliptin (Kombiglyze) Sitagliptin (Januvia) Metformin + Sitagliptin (Janumet) Sitagliptin + Simvastatin (Juvisync) Glucagon-like peptide-1 receptor agonist (GLP-1 RA) with Insulin Albiglutide (Tanzeum) Dulaglutide (Trulicity) Exenatide (Byetta, Bydureon) Rybelsus (Semaglutide) Xultophy (insulin degludec and liraglutide injection) Glargine + Lixisenatide (Soliqua) Liraglutide (Victoza, Saxenda) Lixisenatide (Adlyxin) Semaglutide (Ozempic) Sodium-glucose cotransporter-2 inhibitors (SGLT-2i mono and combi) Canagliflozin (Invokana) Metformin + Canagliflozin (Invokamet) Metformin + Canagliflozin extended-release (Invokamet XR) Dapagliflozin (Farxiga) Empagliflozin (Jardiance) Empagliflozin + Linagliptin (Glyxambi) Metformin + Empagliflozin (Synjardy) Metformin + Empagliflozin extended-release (Synjardy XR) Dapagliflozin + Saxagliptin (Qtern) Metformin + Dapagliflozin extended-release (Xigduo XR) Ertugliflozin (Steglatro) Ertugliflozin + Metformin (Segluromet) Ertugliflozin + Sitagliptin (Steglujan) Insulin

c37922104-02

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

## **ANNEX 3. STUDY COVARIATES**

| N | Category | Variables | Definition |
|---|---|---|---|
| | | Age | - By year<br>- By category (18-54, 55-64, 65-74, 75+) |
| | | Gender | - Male, Female |
| | | Smoking | A 11 1 1 1 1 <b>C</b> 1 : - 4 |
| 1 | Demographics | Alcohol abuse or dependence | All codes could be found in the |
| | | Drug abuse or dependence | following excel file: |
| | | Overweight | <u> </u> |
| | | Obesity | X III |
| | | Calendar quarter of cohort entry | 1245-0201%20codes<br> |
| | | Calendar year of cohort entry | - %20part%201_03022 |
| | Comorbidity | Elixhauser comorbidity index | - <u>R14-4775</u> |
| 2 | indexes | Charlson comorbidity index | |
| | | Diabetes retinal problems | |
| | | Diabetic neuropathy | |
| | | Diabetic nephropathy | |
| | | Hypoglycaemia | |
| | | Hyperglycaemia | |
| | | Disorders of fluid electrolyte and | - Diabetic retinopathy, |
| | | acid-base balance | diabetes with other |
| | | Diabetic ketoacidosis | ophthalmic manifestations, |
| | | Hyperosmolar hyperglycemic | Retinal detachment, |
| | | nonketotic syndrome (HONK) | vitreous hemorrhage, |
| | | Diabetes with peripheral | vitrectomy, retinal laser |
| | | circulatory disorders | coagulation therapy. Codes |
| | Diabetes<br>specific<br>complications | Diabetic foot | presented in the following excel file: |
| 3 | | Gangrene | excel file. |
| | | Lower extremity amputation | |
| | | (lower extremity amputation | X≡ |
| | | diagnosis code, lower extremity | 1245-0201%20codes |
| | | amputation procedure code (ICD), | %20part%201_03022 |
| | | lower extremity amputation | |
| | | procedure code (CPT).) | _ |
| | | Osteomyelitis | _ |
| | | Skin infections | 4 |
| | | Erectile dysfunction | |
| | | Diabetes with unspecified | |
| | | complication | 4 |
| | | Diabetes mellitus without mention | |
| | | of complications | |


| P | roprietary confidential info | ormation © 2022 Boehringer Ingelheim International Gmb | H or one or more of its affiliated companies |
|---|---|---|---|
| | | Hypertension | |
| | | Hyperlipidaemia | |
| | | Myocardial infarction (Acute MI | |
| | | and old MI) | |
| | | Angina (ACS/unstable angina, | |
| | | stable angina) | |
| | | Coronary atherosclerosis and other | |
| | | forms of chronic ischemic heart | |
| | | disease | |
| | | Cardiac procedures (Previous | |
| | | cardiac procedure (CABG or | |
| | | PTCA or Stent)) | <ul> <li>Codes presented in the</li> </ul> |
| | | Ischemic stroke (w and w/o | following excel file: |
| | | mention of cerebral infarction) | - |
| | | Hemorrhagic stroke | |
| | | TIA | X = |
| | | Cerebrovascular disease (Other | 1245-0201%20codes |
| | | cerebrovascular disease, late | %20part%202_03022 |
| | | effects of cerebrovascular disease, | |
| | | Cerebrovascular procedure) | x ≣ |
| | General | Heart failure (CHF) | 1245-0201%20Code |
| 4 | medical | Peripheral Vascular disease or | s%20part%203_0304 |
| | history | PVD surgery | • |
| | , | Atrial fibrillation | |
| | | Other cardiac dysrhythmia Cardiac conduction disorders | X≡ |
| | | Other CVD | 1245-0201%20codes |
| | | COPD | %20part%205_04162 |
| | | Asthma | |
| | | Obstructive sleep apnoea | |
| | | Renal | |
| | | Osteoarthritis | |
| | | Rheumatoid arthritis | |
| | | Dorsopathies | |
| | | Fractures | |
| | | Falls | |
| | | Osteoporosis | |
| | | Hypothyroidism | |
| | | Hyperthyroidism | |
| | | Other disorders of thyroid gland | |
| | | Depression | |
| | | Anxiety | |
| | | Sleep disorders | |
| | | 1 | |
| | | Neoplasms | |

c37922104-02

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)


| Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies | | |
|---|---|---|
| | | Human immunodeficiency virus |
| | | infection |
| | | Ulcerative colitis |
| | | Crohn's disease |
| | | Gastroesophageal reflux disease |
| | | Gastrointestinal haemorrhage |
| 5 | Use of insulin | |
| 6 | Use of other oral hypoglycaemic agents | |
| 7 | Use of drug(s) associated with acute pancreatitis * | α-methyldopa, azodisalicylate, bezafibrate, cannabis, carbimazole, codeine, cytosine, arabinoside, dapsone, enalapril, furosemide, isoniazid, mesalamine, metronidazole, pentamidine, pravastatin, procainamide, pyritonol, simvastatin, stibogluconate, sulfamethoxazole, sulinda, tetracycline, valproic acid, all trans-retinoic acid, amiodarone, azathioprine, clomiphene, dexamethasone, ifosfamide, lamivudine, losartan, lynesterol/methoxyethinylestradiol, Mercaptopurine, meglumine, methimazole, nelfinavir, norethindronate/mestranol, omeprazole, premarin, sulfamethazole, trimethoprimsulfamethazole, acetaminophen, chlorthiazide, clozapine, didanosine, erythromycin, estrogen, L-asparaginase, pegasparagase, propofol, tamoxifen, azathioprine, sulfonamides, tetracyclines, alphamethyldopa |
| 8 | Use of any other medications not mentioned above | <ul> <li>Agents acting on the reninangiotensin system</li> <li>Antibacterials for systemic use</li> <li>Antidepressants</li> </ul> |


| Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies | | | |
|---|---|---|---|
| | | <ul> <li>Antiepileptics</li> </ul> | |
| | | <ul> <li>Antiinflammatory and</li> </ul> | |
| | | antirheumatic products | |
| | | <ul> <li>Antineoplastic agents</li> </ul> | |
| | | <ul> <li>Antipsoriatics</li> </ul> | |
| | | <ul> <li>Antithrombotic agents</li> </ul> | |
| | | <ul> <li>Beta-blocking agents</li> </ul> | |
| | | <ul> <li>Calcium channel blockers</li> </ul> | |
| | | <ul> <li>Diuretics</li> </ul> | |
| | | <ul> <li>Drugs for acid-related</li> </ul> | |
| | | disorders | |
| | | <ul> <li>Drugs for obstructive</li> </ul> | |
| | | airway diseases | |
| | | <ul> <li>Immunosuppressants</li> </ul> | |
| | | <ul> <li>Lipid-modifying agents</li> </ul> | |
| | | • Opioids | |
| | | <ul> <li>Psycholeptics</li> </ul> | |
| | | <ul> <li>Psychostimulants, agents</li> </ul> | |
| | | used for ADHD, and | |
| | | nootropics | |
| | | Abdominal surgery | |
| | History of acute pancreatitis risk factors | • Alcoholism | |
| | | • Cystic fibrosis | |
| | | • Gallstones and other gallbladder and biliary tract | Codes are listed in the |
| | | disorders | following excel file: |
| | | <ul> <li>High calcium levels in the</li> </ul> | |
| 9 | | blood (hypercalcemia) | x ≡ |
| | | Hyperparathyroidism | 1245-0201%20Code |
| | | Hypertriglyceridemia | s%20part%204%20-% |
| | | • Infection | |
| | | • Injury to the abdomen | |
| | | • Lupus | |
| | | • Liver disease | |
| | | <ul> <li>Pancreatic disease</li> </ul> | |
| | Lab test results | • amylase (U/L); | |
| | | • lipase (U/L); | |
| | | • white cell count (G/L); | |
| | | <ul> <li>red cell count (T/L);</li> </ul> | |
| 10 | (when | <ul> <li>haemoglobin (g/L);</li> </ul> | |
| | available) | <ul><li>haematocrit (%);</li></ul> | |
| | | <ul> <li>thrombocyte (G/L);</li> </ul> | |
| | | • C-reactive protein (mg/L); | |
| | | <ul> <li>creatinine (μmol/L),</li> </ul> | |

c37922104-02

Statistical and Epidemiological Analysis Plan (SEAP) for Non-Interventional Studies (NIS)


| Pr | Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies | |
|---|---|---|
| | | carbamid (mmol/L); serum |
| | | bilirubin (μmol/L); |
| | | • GGT (mmol/L); |
| | | • GOT (mmol/L); |
| | | • GPT (mmol/L); |
| | | • ALP (mmol/L); |
| | | • uric acid (mmol/L); |
| | | • cholesterol (HDL, LDL) |
| | | (mmol/L); triglycerides |
| | | (mmol/L); |
| | | • serum protein (g/L); |
| | | • albumin (g/L)., |
| | | C-peptide (pmol/L); |
| | | • HgbA1C (%); |
| | | OGTT test glucose |
| | | (mmol/L) and insulin level |
| | | (pmol/L) at 0, 60 and |
| | | 120min [add reference]. |
| | | • HbA1c (%) |
| | | • LDL level (mg/dl) |
| | | HDL level (mg/dl) |
| | | Total cholesterol (mg/dl) |
| | | Triglyceride level (mg/dl) |
| | | • Creatinine (mg/dl) |
| | | BUN (mg/dl) |
| | | • BNP |
| | | NT-proBNP |
| | | • Lipase |
| 11 | Procedures | Abdominal ultrasound |


Proprietary confidential information © 2022 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### ANNEX 4. REVIEWERS AND APPROVAL SIGNATURES

The NIS SEAP must be sent for review to the following individuals **prior to approval**.

| Reviewer | NIS involving BI<br>product(s) | NIS not involving BI product(s) | |
|---|---|---|---|
| | | Global NIS | Local NIS |
| NIS Lead | X | X | X |
| Global TM Epi* | X | X | X |
| NIS Data Manager | X | X | X |
| TSTAT<br>(for NISnd only) | Х | X | X |
| RWE CoE | X | X | |

<sup>\*</sup> When BI NIS lead is not TM Epi

Study Title: Statistical and Epidemiological Analysis Plan (SEAP) for Post-authorization safety study (PASS) to assess the risk of acute pancreatitis in type 2 diabetes mellitus (T2DM) patients newly initiating empagliflozin compared to other oral non-incretin/non-sodium glucose co-transporter-2 inhibitors (SGLT2)-based hypoglycemic agents – Version 1.0

**Study Number: 1245-0201** 

**Protocol Version:** Version 1.0

I herewith certify that I agree to the content of the study SEAP and to all documents referenced in the study SEAP.

| Position: NIS | Name/Date:<br>Jul 2021 | / 23 | Signature: |
|---|---|---|---|
| Position: TM BDS | Name/Date: | / dd mmm yyyy> | Signature: |
| Position: Global<br>TM Epi | Name/Date:<br>ddmmmyyyy | | Signature: |
| Position: NIS Data | Name/Date: | | Signature: |
| Position: | Name/Date: | | Signature: |